CLINICAL TRIAL: NCT07370935
Title: The Relationship Between Trunk Stability, Balance, Mobility, Upper Limb Performance, and Fatigue in Minimally to Moderately Disabled People With Multiple Sclerosis
Brief Title: Trunk Stability, Balance, and Fatigue in Minimally to Moderately Disabled People With Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Cappadocia University (Other)
Responsible Party: Principal Investigator, Tansu Kus, Assistant Professor, Cappadocia University
Other Study IDs: 25.12
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; balance; mobility; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurements — No intervention. Participants will be assessed observationally for trunk stability, balance, mobility, upper limb performance, and fatigue using standardized clinical tests.

SUMMARY:
The goal of this observational study is to investigate the relationship between trunk stability and balance, mobility, upper limb performance, and fatigue in people with multiple sclerosis (MS) with minimal to moderate disability levels.

The main questions it aims to answer are:

1. Is trunk stability associated with balance, mobility, upper limb performance, and fatigue in people with multiple sclerosis with minimal to moderate disability?
2. Do balance, mobility, upper limb performance, and fatigue differ between minimally and moderately disabled people with multiple sclerosis?

Participants with a diagnosis of multiple sclerosis and Expanded Disability Status Scale (EDSS) scores ≤2 (minimally disabled) and 2.5-4 (moderately disabled) will be included in the study.

Participants will undergo standardized clinical assessments to evaluate trunk stability, balance, mobility, upper limb performance, and fatigue during a single assessment session. No intervention will be applied as part of the study, and all measurements will reflect participants' current functional status.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of multiple sclerosis was confirmed by a neurologist.
* Expanded Disability Status Scale (EDSS) score between 0 and 4
* Age between 18 and 65 years
* Accepting participation in the study voluntarily

Exclusion Criteria:

* An MS attack within the last three months
* Pregnancy
* Presence of cardiovascular, pulmonary, or orthopedic conditions that would prevent participation in exercise
* A disease that can affect the immune system, such as infection or cancer
* Additional neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will consist of adult men and women aged 18-65 years with a confirmed diagnosis of multiple sclerosis living in Ankara.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
The Prone Bridge Test | Single assessment at the time of enrollment
  The prone bridge test was used to assess core muscle endurance. In this test, the individuals were asked to raise their bodies in a prone position, supporting themselves on their forearms and toes with their elbows flexed, maintaining this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was repeated twice, and the longer duration was recorded.
The Side-bridge Test | Single assessment at the time of enrollment
  The side-bridge test was used to assess core muscle endurance. The individuals were positioned in a straight line, lying on their left or right side with their legs fully extended. The individuals were asked to lift their body on forearms and toes, and maintain this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was performed twice, and the longer duration was recorded.
The Trunk Flexor Test | Single assessment at the time of enrollment
  The trunk flexor test was used to assess core muscle endurance. The individuals were positioned in a sit-up position with their back resting against a wedge angled at 60° from the floor. After the wedge was removed, they were asked to maintain this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was repeated twice, and the longer duration was recorded.
The Biering-Sorensen Test | Single assessment at the time of enrollment
  The Biering-Sorensen test was used to assess core muscle endurance. In this test, the individuals were asked to lie prone on a workout bench, aligning their anterior superior iliac spine with the edge of the bench, allowing the upper body to extend over the edge. An assisting partner secured the individuals' knees, hips, and pelvis. The individuals were instructed to fold their arms across their chest and to hold this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was performed twice, and the longer duration was recorded.
The Sit-ups Test | Single assessment at the time of enrollment
  The sit-ups test was used to assess core muscle strength. The test began when the individuals were instructed to ''go'', and they were asked to lift their upper body off the floor, raising the lower corner of the scapula. The score was recorded as the number of repetitions completed in 30 seconds. In the study, the test was performed twice, and the highest number of repetitions was recorded.
The Modified Push-ups Test | Single assessment at the time of enrollment
  The modified push-ups test was used to assess core muscle strength. The individuals were positioned on their hands and knees with hands shoulder-width apart and elbows fully extended. They dropped their hips and moved their hands forward until they created a straight line and a straight back from the knees to the hips to the shoulders. During the test, the individuals were asked to maintain this straight position while lowering their upper body until their elbows were bent to 90°, then pushing back up to the starting position. The score was recorded as the number of repetitions completed in 30 seconds. In the study, the test was performed twice, and the highest number of repetitions was recorded.
The Postural Stability Test | Single assessment at the time of enrollment
  The Postural Stability Test was assessed with The Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). The test evaluates static balance by assessing the individual's ability to maintain their center of gravity over the support surface while standing. During the test, the individuals were asked to stand as still as possible. The test duration was 30 seconds and a total stability index score was calculated. The stability index scores range from 0 to 4, with lower scores indicating good postural stability.
The Limits of Stability Test | Single assessment at the time of enrollment
  The Limits of Stability Test was assessed with The Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). During the test, the individuals were asked to move their bodies toward target points displayed on the screen without lifting their feet and then return to the center point. During this movement, they were instructed to move as quickly and accurately as possible. The test results in a total percentage score. A lower score indicates decreased stability limits.
The Modified Sensory Organization Test | Single assessment at the time of enrollment
  The Modified Sensory Organization Test (MSOT) was assessed with the Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). In the test, by selectively disrupting visual and somatosensory inputs, it is determined which sensory inputs the individual relies on the most to maintain postural stability. The MSOT was performed under four conditions in the study: eyes open on a firm surface, eyes closed on a firm surface, eyes open on a soft surface, and eyes closed on a soft surface. The individuals were instructed to maintain their balance in all conditions. The test duration was 30 seconds for each condition. The sway index scores were calculated at the end of the test. The sway index scores range from 0 to 4, with lower sway index scores indicating decreased postural sway.
The Activities-specific Balance Confidence Scale | Single assessment at the time of enrollment
  The Activities-specific Balance Confidence Scale (ABC) evaluates balance confidence in daily living activities and includes 16 activities related to balance. Participants were asked to rate their perceived safety while performing these activities and their perceived risk of falling on a scale from 0 (completely unsafe) to 100 (completely safe). The total score is calculated by dividing the score by 16 and ranges from 0 to 100. Scores closer to zero indicate greater balance impairment and a higher risk of falls.
The 6-Minute Walk Test | Single assessment at the time of enrollment
  Walking performance and functional exercise capacity were assessed using the Six-Minute Walk Test (6-MWT). Participants were instructed to walk at the highest speed they felt safe in a 30-meter straight pathway for six minutes. The score was the total walking distance in meters at the end of the test.
The Timed Up and Go Test | Single assessment at the time of enrollment
  Functional mobility was assessed by the Timed Up and Go Test (TUG). During the test, the individuals were asked to get up from the chair, walk 3 meters, turn around, walk back to the chair, and sit down. The score was the total time in seconds to complete the task. In the study, the test was repeated three times, and the average time was recorded.
The Five Times Sit-to-Stand Test | Single assessment at the time of enrollment
  Lower extremity functional muscle strength was assessed by the Five Times Sit-to-Stand Test. The individuals were seated in a standard chair with arm support of 43-45 cm height, with their arms crossed on their chests. When the command "Start" was given, individuals were asked to stand up as quickly as possible and sit down and stand up 5 times. The score was the total time in seconds to complete the task. In the study, the test was repeated twice and the shortest time was recorded.

SECONDARY OUTCOMES:
The Nine-Hole Peg Test | Single assessment at the time of enrollment
  Upper extremity performance was assessed using the Nine-Hole Peg Test (9-HPT). The 9-HPT consists of a pegboard with 9 holes and 9 wooden pegs. Individuals were asked to place and remove all 9 pegs one at a time as fast as possible. The score was the total time in seconds to complete the task. In the study, the test was repeated twice for each extremity, and the average time was recorded for each side.
The Fatigue Severity Scale | Single assessment at the time of enrollment
  The Fatigue Severity Scale (FSS) assesses the severity of fatigue in the last month. It consists of 9 items, and the items are scored from 1 (strongly disagree) to 7 (strongly agree). The mean of the nine item scores is used as the FSS score. The scores that can be obtained from the test are between 1 and 7, and high scores indicate the presence of fatigue.
The Fatigue Impact Scale | Single assessment at the time of enrollment
  The Fatigue Impact Scale (FIS) assesses the impact of fatigue on physical, cognitive, and psychosocial functions in the last four weeks. It consists of 40 questions, with responses ranging from 0 (no problem) to 4 (extreme problem). The scores that can be obtained from the test are between 0 and 160, and high scores indicate a greater fatigue effect.